CLINICAL TRIAL: NCT05503095
Title: PCSK9 Polymorphism and Risk of Mechanical Complications Following Acute Myocardial Infarction
Brief Title: PCSK9 Polymorphism and Risk of Cardiac Rupture
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: IT-VA-237-2021
Record Dates: First submitted 2022-08-09; First posted 2022-08-16 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Post-Infarction Heart Rupture; Gene Polymorphism
Keywords: PCSK9; Cardiac rupture
MeSH Terms: conditions — Heart Rupture, Post-Infarction; Heart Rupture | interventions — Genetic Testing

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients who develop cardiac rupture following acute myocardial infarction
  Interventions: Genetic: Genetic analysis for PCSK9 polymorphisms
- patients with acute ST-elevation myocardial infarction not complicated by cardiac rupture
  Interventions: Genetic: Genetic analysis for PCSK9 polymorphisms

INTERVENTIONS:
Genetic: Genetic analysis for PCSK9 polymorphisms — Determination of PCSK9 gene polymorphism and serum PCSK9 concentration

SUMMARY:
Protein convertase subtilisin/kexin type 9 (PCSK9) plays a regulatory role in cholesterol homeostasis by promoting low-density lipoprotein receptor (LDLr) degradation. Although the vast majority of the studies have focused on the role of PCSK9 in LDLr expression in the liver, an increasing body of evidence suggests that PCSK9 gene is also present in extra-hepatic tissues. A recent publication showed for the first time that PCSK9 is expressed in the ischemic heart and the expression is highest in the zone bordering the infarcted areas. Furthermore, the expression of PCSK9 is maximal early, at 1 week of ischemia.

Mechanical complications (or cardiac ruptures) are uncommon but potentially lethal sequelae of acute myocardium infarction (AMI) and are commonly associated with early mortality without appropriate surgical intervention. It's unknown why some patients develop these devasting complications following AMI, while others not. Interestingly, studies have shown that post-infarction cardiac rupture affect the border zone between the ischemic and normal area and occur within the first 3 to 5 days after AMI.

Based on the aforementioned observations, it's likely to assume a relationship between PCSK9 expression and the development of post-AMI cardiac rupture. Therefore, the main purpose of the this project is to study the PCSK9 gene polymorphism and its association with cardiac rupture. Investigators hypothesize that PCSK9 expression/secretion and development of post-AMI cardiac rupture may be a part of the dynamic changes at cellular levels occurring in the ischemic heart of genetically predisposed patients.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of acute myocardial infarction with ST sopra-elevation (control group)
* clinical diagnosis of acute myocardial infarction complicated by cardiac rupture

Exclusion Criteria:

* absence of coronary artery disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who develop cardiac rupture following acute myocardial infarction (case group) and patients with acute ST-elevation myocardial infarction not complicated by cardiac rupture (control group)
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
PCSK9 gene polymorphism | up to 1 year
  PCSK9 gene polymorphism (studied at patient admission and recovery for acute myocardial infarction)

CONTACTS AND LOCATIONS:
Locations (1):
- Matteo Matteucci, Varese, Italy

IPD SHARING:
Plan to Share IPD: Undecided